CLINICAL TRIAL: NCT03159611
Title: Multicenter Double-blind Placebo-controlled Parallel-group Randomized Clinical Trial of Efficacy and Safety of Tenoten for Children Liquid Dosage Form Therapy in Infants With Sequelae of Perinatal Brain Injury
Brief Title: Efficacy and Safety Clinical Trial of Tenoten for Children Liquid Dosage Form Therapy in Infants With Sequelae of Perinatal Brain Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-TD-004
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Results first posted 2019-04-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Sequelae of Perinatal Brain Injury
MeSH Terms: interventions — tenoten

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tenoten for children (Experimental)
  Interventions: Drug: Tenoten for children
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tenoten for children — Oral. 10 drops daily, at the same time in the morning, 15 minutes before feeding.
  Arms: Tenoten for children
Drug: Placebo — Oral. 10 drops daily, at the same time in the morning, 15 minutes before feeding.
  Arms: Placebo

SUMMARY:
Purpose of the study:

* To assess the clinical efficacy of Tenoten for children liquid dosage form therapy (10 oral drops per day for 12 weeks) in Infants with Sequelae of Perinatal Brain Injury (mild-to-moderate cerebral hypoxia-ischaemia and/or mild-to-moderate intracranial haemorrhage).
* To assess the safety of Tenoten for children liquid dosage form therapy (10 oral drops per day for 12 weeks) in Infants with Sequelae of Perinatal Brain Injury (mild-to-moderate cerebral hypoxia-ischaemia and/or mild-to-moderate intracranial haemorrhage).

ELIGIBILITY:
Inclusion Criteria:

1. Full-term infants aged 29 days to 9 months.
2. Diagnosis of Sequelae of Perinatal Brain Injury (mild-to-moderate cerebral hypoxia-ischemia and/or mild-to-moderate intracranial hemorrhage).
3. Total Jurba-Mastyukova score of < 27 (but > 12).
4. Physical development parameters within 25-27 centiles.
5. Neurologist's outpatient observation.
6. Information sheet (informed consent form) for parents/adoptive parents for participation in the clinical study signed by the child's parents/adoptive parents.

Exclusion Criteria:

1. Previously diagnosed lesions, diseases and conditions:

   1.1. Cerebral ischemia (grade III). 1.2. Intraventricular hemorrhage (grade III). 1.3. Metabolic and toxic disorders affecting central nervous system (persistent neonatal hypoglycemia, hyperbilirubinemia associated with elevated indirect bilirubin, and other severe conditions).

   1.4. Intracranial birth injury, focal impairments due to brain injuries (pareses and paralyses).

   1.5. Sequelae of birth injury to spinal cord, cranial nerves and peripheral nervous system (peripheral pareses and paralyses).

   1.6. Different types of hydrocephalus. 1.7. Symptomatic epilepsy and epileptic syndromes. 1.8. Sequelae of perinatal central nervous system (CNS) infectious diseases (injury to CNS caused by neonatal sepsis, encephalitis, meningitis, meningoencephalitis, ventriculitis).

   1.9. Infectious diseases including congenital diseases (cytomegalovirus infection, rubella, herpesvirus or enterovirus infection, toxoplasmosis, syphilis, HIV infection, etc.).

   1.10. Chronic respiratory diseases originating in the perinatal period, including bronchopulmonary dysplasia.

   1.11. Hereditary metabolic diseases including glycogen storage disease (glycogenoses, E74.0), galactose metabolism disorders (galactosemia, Е74.2), other carbohydrate metabolism disorders (Е74), glucosaminoglycan metabolism disorders (mucopolysaccharidoses, Е76), aromatic amino-acid metabolism disorders (phenylketonuria, tyrosinemia, etc, Е70), branched-chain amino-acid and fatty-acid metabolism disorders (maple-syrup-urine disease, Е71), mitochondrial myopathy (G71.3).

   1.12. Neurogenerative diseases including Huntington disease (G10), copper metabolism disorder (Wilson disease, Е83.0).

   1.13. Chromosomal abnormalities. 1.14. Congenital anomalies [malformations] and deformities including congenital anomalies of nervous system and malformations of internal organs.

   1.15. Congenital endocrine diseases (congenital hypothyroidism, hypoparathyroidism, adrenocortical dysfunction).

   1.16. Malignant neoplasm / suspected malignant neoplasm.
2. Acute infectious disease, exacerbation / decompensation of diseases that may prevent the patients' participation in the clinical study.
3. Allergy/intolerance of any of the study treatment medications components.
4. Drug addiction, alcohol use in the volume over 2 alcohol units/day by the subject's parent(s)/adoptive parent(s).
5. Mental disorders of the patient's parent(s)/adoptive parent(s).
6. Participation in other clinical studies for a period prior to and during the course of this trial.
7. Other conditions complicating the subject's participation in the study (cannot make regular medical visits, moving, etc.).
8. Subjects whose parent(s)/adoptive parent(s), from the investigator's point of view, will not follow the study requirements or comply with the dosing regimen.
9. Patients whose parent(s)/adoptive parent(s) are related research staff of the clinical investigative site who are directly involved in the study or is a close relative of the investigator. Close relatives include spouse, parents, children or brothers (sisters) regardless of whether they are biological or adoptive ones.
10. Patients whose parent(s)/adoptive parent(s) is working in OOO "NPF "Materia Medica Holding", i.e. is the company official, temporary contract worker or an appointed official responsible for the study or their close relatives.

Ages: 29 Days to 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 182 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2018-02-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- Russia (10):
  - Federal State Budgetary Educational Institution of Higher Education "Kazan Medical University" of the Ministry of Healthcare of the Russian Federation, Kazan'
  - Pirogov Russian National Research Medical University, Moscow
  - I.M. Sechenov First MSMU, Moscow
  - Moscow Regional Research and Clinical Institute ("MONIKI"), Moscow
  - Municipal Health Care Institution "City Child Health Clinical Polyclinic №5", Perm
  - State budgetary institution of public health of the Samara region "Samara City Children's Clinical Hospital No. 1 named after N.N. Ivanova", Samara
  - LLC "Center for DNA Research", Saratov
  - LLC Nebbiolo, Tomsk
  - Federal State Budgetary Educational Institutionof Higher Education "Yaroslavl State Medical University" of the Ministry of Healthcare of the Russian Federation, Yaroslavl
  - State Budgetary Healthcare Institution of Sverdlovsk Region Children's Clinical Hospital of Rehabilitation The Scientific and Practical Center "Bonum", Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo: Oral. A dose of 10 drops daily, at the same time in the morning, 15 minutes before feeding the child.
  The drops can be diluted in a small amount of room temperature drinking water (1/2 tsp.) before use.
- Tenoten for Children: Tenoten for children: Oral. A dose of 10 drops daily, at the same time in the morning, 15 minutes before feeding the child.
  The drops can be diluted in a small amount of room temperature drinking water (1/2 tsp.) before use.
Period: Overall Study
Arm/Group | Placebo | Tenoten for Children
Started | 95 | 87
Completed | 72 | 72
Not Completed | 23 | 15
Not completed — Did Not Meet Inclusion Criteria | 9 | 5
Not completed — Did Not Meet Exclusion Criteria | 1 | 3
Not completed — Protocol Violation | 7 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Non-compliance with protocol requirement | 3 | 2
Not completed — Inability to perform procedures | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenoten for Children | Placebo | Total
Number analyzed (Participants) | 87 | 95 | 182
Age, Continuous [Mean (Standard Deviation); unit: months] | 5.5 (2.0) | 5.0 (2.3) | 5.2 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 41 | 83
  Male | 45 | 54 | 99
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body length [Mean (Standard Deviation); unit: centimeter] | 63.9 (4.6) | 62.5 (5.3) | 63.2 (5.0)
Head circumference [Mean (Standard Deviation); unit: centimeter] | 42.0 (2.3) | 41.4 (2.7) | 41.7 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With a 4 and More Point Increase of the Total Score According to Jurba-Mastyukova Psychomotor Development Scale by the End of the Treatment
Description: The Jurba-Mastyukova scale is meant to evaluate motor and mental development of 1-12-month-old infants. 10 developmental domains are evaluated every month. The evaluation of each domain is based on a 4-point system (the optimal development equals 3 points, its absence = 0 points). The maximum score is 30 points; 27-29 points are considered as "age-appropriate normal value"; 23-26 points - as "an absolute risk group"; 13-22 points - as "developmental retardation"; below 13 points - as "severe global developmental delay".
Time Frame: in 12 weeks of the treatment
Population: Per Protocol set
Measure: Number; unit: percentage of participants
Arm/Group | Tenoten for Children | Placebo
Number analyzed (Participants) | 72 | 72
percentage of participants | 86.1 | 62.5
Statistical Analysis 1: Comparison: Tenoten for Children vs Placebo; Test type: Superiority; p = 0.002, Fisher Exact

2. Secondary Outcome: Percentage of Patients With Normal Psychomotor Development (≥ 27 Scores on Jurba-Mastyukova Scale) by the End of Treatment Course Compared to Baseline (Time Frame: 0 Weeks, 4 Weeks, 8 Weeks, 12 Weeks)
Description: as for outcome 1
Time Frame: in 12 weeks of the treatment
Population: Per Protocol set
Measure: Number; unit: Percentage of patients
Arm/Group | Tenoten for Children | Placebo
Number analyzed (Participants) | 72 | 72
Percentage of patients
  Week 4 | 45.8 | 34.7
  Week 8 | 79.2 | 66.7
  Week 12 | 93.1 | 81.9
Statistical Analysis 1: Comparison: Tenoten for Children vs Placebo; Test type: Superiority; p = 0.005, Cochran-Mantel-Haenszel

3. Secondary Outcome: Mean Cognitive Adaptive Test/Clinical Linguistic and Auditory Milestone Scale (CAT/CLAMS) Score by the End of the Treatment Course Compared to Baseline (Time Frame: 0 Weeks, 4 Weeks, 8 Weeks, 12 Weeks)
Description: The Clinical Adaptive Test/Clinical Linguistic and Auditory Milestone Scale (CAT/CLAMS) Consists of Three batteries: Clinical adaptive test (CAT), clinical linguistic and auditory milestone scale (CLAMS), and Gross motor (GM). CAT is the visual-motor problem-solving battery; the score on the CAT is based on the child's performance with the administered items. CLAMS is the language battery of the test; the score on the CLAMS is based on the parent's report of language skill attainment. GM evaluates motor skills; the score on the GM is based on the direct observation of a child and examination by the neurologist. The scores from the CAT/CLAMS+GM are expressed as developmental quotients [DQ = (developmental age/chronologic age)*100]. The full-scale CAT/CLAMS+GM DQ (full-scale DQ) is the mean of the CAT DQ, the CLAMS DQ, and GM DQ. Full-scale DQ ≥ 75 is considered as normal value (the child has a normal development).
Time Frame: in 12 weeks of the treatment
Population: Per Protocol set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tenoten for Children | Placebo
Number analyzed (Participants) | 72 | 72
score on a scale
  Week 0 | 86.2 (14.2) | 83.5 (16.9)
  Week 4 | 92.5 (14.1) | 90.6 (12.9)
  Week 8 | 95.4 (10.5) | 94.6 (11.3)
  Week 12 | 97.5 (8.9) | 95.2 (10.3)
Statistical Analysis 1: Comparison: Tenoten for Children vs Placebo; Test type: Superiority; p = 0.50, Mixed Models Analysis

4. Secondary Outcome: Percentage of Patients With Normal Psychomotor Development (CATS/CLAMS + Gross Motor Developmental Quotients Score ≥ 75) by the End of the Treatment Course Compared to Baseline (Time Frame: 0 Weeks, 4 Weeks, 8 Weeks, 12 Weeks)
Description: The Clinical Adaptive Test/Clinical Linguistic and Auditory Milestone Scale (CAT/CLAMS) Consists of Three batteries: Clinical adaptive test (CAT), clinical linguistic and auditory milestone scale (CLAMS), and Gross motor (GM). CAT is the visual-motor problem-solving battery. The score on the CAT is based on the child's performance with the administered items. CLAMS is the language battery of the test. The score on the CLAMS is based on the parent's report of language skill attainment. GM evaluates motor skills. The score on the GM is based on the direct observation of a child and examination by the neurologist. The scores from the CAT/CLAMS+GM are expressed as developmental quotients [DQ = (developmental age/chronologic age)*100]. The full-scale CAT/CLAMS+GM DQ (full-scale DQ) is the mean of the CAT DQ, the CLAMS DQ, and GM DQ. Full-scale DQ ≥ 75 is considered as normal value (the child has a normal development).
Time Frame: in 12 weeks of the treatment
Population: Per Protocol set
Measure: Number; unit: Percentage of patients
Arm/Group | Tenoten for Children | Placebo
Number analyzed (Participants) | 72 | 72
Percentage of patients
  Week 0 | 81.9 | 77.8
  Week 4 | 91.7 | 91.7
  Week 8 | 100 | 97.2
  Week 12 | 100 | 95.8
Statistical Analysis 1: Comparison: Tenoten for Children vs Placebo; Test type: Superiority; p = 0.20, Cochran-Mantel-Haenszel

5. Secondary Outcome: Clinical Global Impression Scale - Efficacy Index (CGI-EI) Score by the End of the Treatment Course.
Description: The Clinical Global Impressions - Efficacy Index (CGI-EI) scale provide an evaluation of the treatment response. CGI-EI takes account of both therapeutic efficacy and treatment-related adverse events and ranges from 0 (marked improvement and no side-effects) and 4 (unchanged or worse and side-effects outweigh the therapeutic effects).
Time Frame: in 12 weeks of the treatment
Population: Per Protocol set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tenoten for Children | Placebo
Number analyzed (Participants) | 72 | 72
score on a scale
  Therapeutic effect | 3.4 (0.6) | 3.2 (0.8)
  Side effect | 1.1 (0.3) | 1.0 (0.1)
  Efficacy Index | 3.2 (0.8) | 3.2 (0.8)
Statistical Analysis 1: Comparison: Tenoten for Children vs Placebo; Test type: Superiority; p = 0.19, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse/Serious adverse events were registered during 12 weeks of therapy.
Description: Adverse/Serious adverse events were registered in patients of the Full Analysis Set (n=182, Safety Population)
Arm/Group | Tenoten for Children | Placebo
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/95
Serious Adverse Events (participants affected / at risk) | 1/87 | 0/95
Other Adverse Events (participants affected / at risk) | 24/87 | 27/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenoten for Children (N=87) | Placebo (N=95)
Acute bronchitis (Infections and infestations) | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenoten for Children (N=87) | Placebo (N=95)
Respiratory tract infection (Infections and infestations) | 11 (14) | 8 (9)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Teething (Gastrointestinal disorders) | 5 (5) | 4 (5)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Hyperoxaluria (Renal and urinary disorders) | 1 (1) | 0 (0)
Eczema weeping (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (3)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 2 (2)
Tracheobronchitis (Infections and infestations) | 0 (0) | 2 (2)
Yawning (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rickets (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT03159611/Prot_SAP_000.pdf